CLINICAL TRIAL: NCT00573729
Title: Pulsed Dye Laser Treatment of Port Wine Stain Birthmarks: Comparison of 577 nm Versus 595 nm Wavelengths
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J.S.Nelson, MD,PhD,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20065401
Record Dates: First submitted 2007-12-06; First posted 2007-12-14 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stains
Keywords: vascular malformation
MeSH Terms: conditions — Hemangioma, Capillary; Vascular Malformations | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsed Dye Laser 577 nm (Experimental): Pulsed Dye Laser Treatment 577 nm treatment of Port Wine Stain Birthmarks
  Interventions: Other: Pulsed Dye Laser 577 nm
- Pulsed Dye Laser 595 nm (Experimental): Pulsed Dye Laser Treatment 595 nm treatment of Port Wine Stain Birthmarks
  Interventions: Other: Pulsed Dye Laser 595 nm

INTERVENTIONS:
Other: Pulsed Dye Laser 577 nm — Comparison of 577 nm Versus 595 nm Wavelengths of Pulsed Dye Laser Treatment of Port Wine Stain Birthmarks
  Other Names: Pulsed Dye Laser Treatment of Port Wine Stain Birthmarks
  Arms: Pulsed Dye Laser 577 nm
Other: Pulsed Dye Laser 595 nm — Comparison of 577 nm Versus 595 nm Wavelengths of Pulsed Dye Laser Treatment of Port Wine Stain Birthmarks
  Other Names: Pulsed Dye Laser Treatment of Port Wine Stain Birthmarks
  Arms: Pulsed Dye Laser 595 nm

SUMMARY:
Port wine stain are a congenital, progressive vascular malformation of human skin. The pulsed dye laser is approved by the Food and Drug Administration for the treatment of choice. However, the degree of port wine stain blanching seen following pulsed dye laser treatment remains variable and unpredictable. If the ultimate standard required is complete lesion blanching, the average success rate is below 10%, even after undergoing numerous pulsed dye laser treatments. Moreover, less than 50% of patients achieve 50% fading of their Port wine stain in response to pulsed dye laser therapy.

DETAILED DESCRIPTION:
The researchers' specific aim is to determine whether the use of the pulsed dye laser operating at a wavelength of 577 nm will improve therapeutic outcome as compared to a pulsed dye laser operating at 595 nm.

The researcher can treat port wine stain treated using a pulsed dye laser operating at a wavelength of 577 nm and the other half at a wavelength of 595 nm. The researcher can determine that the 577 nm pulsed dye laser improved port wine stain blanching responses more than the areas treated with 595 nm.

The degree of port wine stain blanching which will determine by visible reflectance spectroscopy skin imaging device measurements. Post-treatment blanching responses can compare with pre-treatment measurements of port wine stain fractional blood volume.

ELIGIBILITY:
Inclusion Criteria:

* Port Wine Stain suitable for comparison testing
* Age > 6 months of age; minor will be accompanied in the room by parents or guardians during laser treatment
* Apparent good health as documented by medical history
* Ability to understand and carry out subject instructions

Exclusion Criteria:

* History of photodermatoses or skin cancer
* Any therapy within the previous two months to the proposed Port Wine Stain treatment sites
* Inability to understand and carry out instructions

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Improvement in blanching for the 577 nm Pulsed Dye Laser therapy in comparison with 595 nm | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S Nelson, M.D., Ph.D., Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute,University of California,Irvine, Irvine, California, United States